CLINICAL TRIAL: NCT06168812
Title: Sulfonylurea Safety and Effectiveness (SUSS) for Patients With Hyperglycemia and Pancreatic Ductal Adenocarcinoma: A Pragmatic Clinical Trial and Accompanying Retrospective Revie
Brief Title: A Study of Glipizide to Treat High Blood Sugar in People With Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-318
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Pancreatic Carcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer Metastatic; Metastatic Pancreatic Cancer; Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Cancer; Pancreatic Carcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer Metastatic; Metastatic Pancreatic Cancer; Metastatic Pancreatic Ductal Adenocarcinoma; Glipizide; Memorial Sloan Kettering Cancer Center; 23-318
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Glipizide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants in this cohort will receive glipizide for up to 4 months and participate in continuous glucose monitoring for as long as they are receiving the drug.
  Interventions: Drug: Glipizide
- Cohort 2a (No Intervention): Participants in this cohort will include people who have received various types of treatment for their hyperglycemia and pancreatic cancer. People's medical records will be reviewed to compare the effects of glipizide with the effects of other standard medications used to treat hyperglycemia.
- Cohort 2b (No Intervention): Participants in this cohort will complete a questionnaire about their use of hyperglycemia medications. Participants from Cohort 2a will take part in this group.

INTERVENTIONS:
Drug: Glipizide — The therapeutic intervention in this study involves the sulfonylurea glipizide in ER formulation.
  Other Names: sulfonylurea glipizide; Glucotrol
  Arms: Cohort 1

SUMMARY:
The purpose of this study is to find out how effective and safe glipizide is for lowering blood sugar in people with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* Age ≥18 years
* Biopsy-proven PDAC
* Radiological evidence and clinical assessment that patient has active disease (local, locally advanced, or metastatic)
* Willing and able to comply with the requirements of the protocol
* Willing to use their bluetooth-enabled wifi or cellular mobile device
* Hemoglobin A1c (HbA1c) > 7%, or fructosamine > 287 mg/dL, or random glucose > 180 mg/dL, or strong clinical suspicion that patient has hyperglycemia, making it reasonable to expect their mean daily glucose is ≥154 mg/dL
* Eastern Cooperative Oncology Group performance status ≤2
* BMI <30 kg/m2

Cohort 2a

* Age ≥18 years
* Biopsy-proven PDAC
* Radiological evidence and clinical assessment that patient has active disease (local, locally advanced, or metastatic pancreatic cancer)
* Clinical diagnosis of diabetes mellitus
* Active care at MSK (defined as at least 1 physician or APP encounter every 3 months) for PDAC during the period from which data were recorded in the electronic medical record (in this retrospective study patients need not be under active care at the time the research is conducted)
* At least 1 electronic prescription for a sulfonylurea (glipizide, glimepiride, or glyburide) or metformin
* Three-month baseline period before metformin or sulfonylurea initiation in which the participant does not receive either drug class or insulin
* Body weight recorded within 3 months before start of metformin or a sulfonylurea

Cohort 2b

* Age ≥18 years
* Biopsy-proven PDAC
* Radiological evidence and clinical assessment that patient has active disease (local, locally advanced, or metastatic)
* Active care at MSK (defined as at least 1 physician or APP encounter every 3 months) for PDAC during the period of data collection
* Apparent current use based on chart review of metformin (but not sulfonylurea); sulfonylurea (but not metformin); or neither drug

Exclusion Criteria:

Cohort 1

* Use during the past month of any antidiabetic medication other than metformin at home (sporadic use [fewer than 1 of 7 days during the past month] is permitted)
* Changes in metformin dose in the past month
* History of sulfonylurea intolerance or allergy
* History of severe hypoglycemia (hypoglycemia requiring emergency medical assistance, emergency room or urgent care visit, or hospital admission)
* AST or ALT >3 x upper limit of normal
* Glomerular filtration rate <30 mL/min/1.73m2
* Daily chronic use of any dose of corticosteroids (as distinct from intermittent exposure to steroids as part of cyclic chemotherapy)
* Inability to wear CGM

Cohort 2a

* Greater than trace ascites documented on imaging or physical exam

Cohort 2b

* Greater than trace ascites documented on imaging or physical exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Change in mean interstitial glucose level for Cohort 1 participants before and after initiation of glipizide | 48 hours after glipizide initiation
  The mean value measured over a 48-h period before initiation of glipizide will be compared with the mean value measured over a 48-h period after glipizide initiation for participants in Cohort 1

CONTACTS AND LOCATIONS:
Overall Officials: James Flory, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication.
Access Criteria: The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required.
URL: https://www.mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org